CLINICAL TRIAL: NCT07379684
Title: A Phase 1 Study to Assess Safety and Tolerability of Amicidin-β Topical Solution in Adult Patients Undergoing Interventional Management of a Surgical or Traumatic Wound Infection
Brief Title: A Study of Amicidin-β Topical Solution for Patients With Surgical or Traumatic Wound Infections
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Macro Biologics, Inc. (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency); Novo Nordisk Foundation (NNF23SA0088536) (Unknown); Global Antimicrobial Resistance Innovation Fund-(GAMRIF) (Unknown); US NIH Grant/Contract Award Number: HHS/BARDA OTA No. 75A50122C00028 (Unknown); Wellcome Trust 224842/Z/21/Z (Unknown); Germany's Federal Ministry of Education and Research (BMBF) Agreement Dated 1/30/23 (Unknown); UK Secretary of State for Health and Social Care ("DHSC"), Agreement dated 02/28/2023 (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BETA-TS-001; 224842/Z/21/Z (Other Grant/Funding Number: Wellcome Trust); Agreement dated 02/28/2023 (Other Grant/Funding Number: UK Secretary of State for Health and Social Care ("DHSC")); Agreement Dated 01/30/2023 (Other Grant/Funding Number: Germany's Federal Ministry of Education and Research (BMBF))
Record Dates: First submitted 2026-01-06; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Surgical Wound Infection; Traumatic Wound Infection
Keywords: Surgical wound infection; Traumatic wound infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SOC + Amicidin-β topical solution - 15 mL (Experimental): In addition to Standard of Care (SOC), patients will receive Amicidin-β topical solution - 15 mL immediately prior to wound closure/dressing, with rinsing out with saline.
  Interventions: Drug: Amicidin-β topical solution - 15 mL; Drug: Standard of Care (SOC)
- SOC + Amicidin-β topical solution - 50 mL - Scheme 1 (Experimental): In addition to Standard of Care (SOC), patients will be receive Amicidin-β topical solution - 50 mL immediately prior to wound closure/dressing, with rinsing out with saline
  Interventions: Drug: Amicidin-β topical solution - 50 mL; Drug: Standard of Care (SOC)
- SOC + Amicidin-β topical solution - 50 mL - Scheme 2 (Experimental): In addition to Standard of Care (SOC), patients will be receive Amicidin-β topical solution - 50 mL immediately prior to wound closure/dressing, without rinsing out with saline
  Interventions: Drug: Amicidin-β topical solution - 50 mL; Drug: Standard of Care (SOC)
- SOC (Active Comparator): Patients will receive Standard of Care (SOC) only
  Interventions: Drug: Standard of Care (SOC)

INTERVENTIONS:
Drug: Amicidin-β topical solution - 15 mL — Amicidin-β topical solution for local administration - 15 mL
  Arms: SOC + Amicidin-β topical solution - 15 mL
Drug: Amicidin-β topical solution - 50 mL — Amicidin-β topical solution for local administration - 50 mL
  Arms: SOC + Amicidin-β topical solution - 50 mL - Scheme 1; SOC + Amicidin-β topical solution - 50 mL - Scheme 2
Drug: Standard of Care (SOC) — Per institutional Standard Of Care

SUMMARY:
The goal of this Phase 1 clinical trial is to learn about the safety profile of Amicidin-β topical solution applied directly into infected surgical or traumatic wounds during a surgical procedure. The main questions it aims to answer are:

1. Is Amicidin-β topical solution safe to test in larger clinical trials?
2. Is Amicidin-β topical solution absorbed into the bloodstream from local wound application?
3. Is Amicidin-β topical solution easy for the surgeon to use? Participants will receive either standard of care alone, or standard of care with intrawound Amicidin-β topical solution for the management of their wound infection. Researchers will compare these two groups (standard of care alone to standard of care with Amicidin-β topical solution) to see if there are any study drug-related adverse effects.

DETAILED DESCRIPTION:
This is a Standard of Care (SOC)- controlled study of approximately 44 patients divided into three sequential cohorts of 8, 12, and 24 patients. Within each sequential cohort, patients will be randomized to SOC only or to SOC plus Amicidin-β topical solution in a 1:3 ratio.

ELIGIBILITY:
Main Inclusion Criteria:

* Body Mass Index between 18.5 kg/square meter and 39.9kg/square meter
* Surgical or traumatic wound determined by the Investigator to be infected within 30 days of surgery or trauma, with longest dimension between 3 and 15 cm. The diagnosis should include one or more of the following signs or symptoms:

  * Purulent drainage
  * Erythema
  * Surrounding induration
  * Fever or localized heat surrounding the wound
  * Reported localized pain or localized tenderness on examination
* Infected surgical or traumatic wound that is determined by the Investigator to required an interventional procedure, such as incision, drainage, irrigation, and/or debridement.
* If female of childbearing potential, must have been practicing an acceptable method of birth control as judged by the Investigator for at least one month prior to enrollment.
* Females of childbearing potential must agree that for the entire duration of the study (about 30 days), they will either practice true abstinence consistent with their preferred and usual lifestyle, or use double contraceptive methods.

Main Exclusion Criteria:

Patients with any of the following will be excluded:

* Surgical or traumatic wound associated with surrounding cellulitis extending ≥10 cm from the wound edge
* Necrotizing fasciitis or gangrenous ulcer
* Multiple surgical or traumatic wound infections at different sites
* Surgical or traumatic wound infection overlying unhealed bone fracture
* Surgical or traumatic wound infection with open peritoneal cavity
* Surgical or traumatic wound infection extending to an organ space
* Surgical or traumatic wound infection with or adjacent to implanted surgical hardware. Note: surgical drains and packing are permitted
* Surgical or traumatic wound infection involving head and neck
* Surgical or traumatic wound infection involving burn injury
* Suspected or confirmed osteomyelitis or septic arthritis
* Surgical or traumatic wound infection known or suspected to be caused by fungal or mycobacterial organisms
* Wound with diagnosis of neuropathic or diabetic foot ulcer or a previous diagnosis of moderate to severe chronic venous insufficiency of a lower extremity in patients with an infected surgical to traumatic wound of the lower extremity
* Wound due to malignancy
* Antibiotic therapy for an infection other than the surgical or traumatic wound infection
* Patient requires supplemental O2 or mechanical ventilation
* Pulse Oximetry (SpO2) reading of ≤ 92% on room air (confirmed by two additional readings ≤92% over 15 min). At geographic locations of high altitude, a lower SpO2 limit (e.g., ≤ 91%) may be used at Investigator's discretion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-10-28 (Estimated); Study Completion 2026-10-28 (Estimated)

PRIMARY OUTCOMES:
Overall comparison of treatment emergent adverse events (TEAES) of combined SOC + Amicidin-β topical solution recipients to SOC only recipients across 3 cohorts. | From Day 1 to Day 30

SECONDARY OUTCOMES:
Number of participants with Treatment Emergent Adverse Events (TEAEs) by severity according to the study protocol. | From Day 1 to Day 30
Measurement of systemic absorption of Amicidin-β recipients. | From Day 1 to Day 3
  Systemic absorption will be assessed by single molecule array (Simoa) immunoassay measurements of patient plasma.

IPD SHARING:
Plan to Share IPD: No